CLINICAL TRIAL: NCT06258161
Title: Functional Reach Test as a Clinical Tool for Assessing Postural Balance Limits Among Adult Spinal Deformity Patients
Brief Title: Effect of Adult Spinal Deformity Surgery on Functional Reach
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Scoliosis Research Society (Other)
Responsible Party: Principal Investigator, Damon Mar, PhD, Research Instructor, University of Kansas Medical Center
Other Study IDs: STUDY00150790
Record Dates: First submitted 2024-01-18; First posted 2024-02-14 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Scoliosis; Scoliosis Kyphosis
Keywords: Balance
MeSH Terms: conditions — Scoliosis | interventions — Spinal Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult spinal deformity surgery patients: Adults diagnosed with spinal deformity and who are undergoing spinal realignment fusion surgery.
  Interventions: Procedure: Spinal Fusion
- Asymptomatic adult controls: Adults with no history of spinal deformity or previous spinal fusions.
  Interventions: Other: No intervention

INTERVENTIONS:
Procedure: Spinal Fusion — Realignment and fusion of adult spinal deformity
  Groups: Adult spinal deformity surgery patients
Other: No intervention — No intervention for control group.
  Groups: Asymptomatic adult controls

SUMMARY:
Adult spinal deformity (ASD) is a common spinal condition that often impacts an individual's ability to stand and maintain an upright posture. Poor balance often limits an individual's ability to perform basic activities of daily life (ADL) and can lead to disability. Current considerations of correcting ASD to improve balance focus on the amount of sway that one exhibits during normal standing. However, current tests do not provide insight into the limits of balance during normal ADL.

The goal of this research is to develop a new balance assessment that includes a functional reach test (FRT) to provide numerical data on the limits of one's ability to maintain balance. The study will include both ASD patients and matched healthy adults and will compare postural sway measures between them. Wearable motion tracking sensors and a force plate will be used to monitor body movement and changes in the center of pressure under foot during normal standing and during a FRT. Data from this study will inform spine surgeons of ASD patient's risk of balance loss in daily life and enable further research on the effects of surgical techniques to restore balance among ASD surgery patients.

DETAILED DESCRIPTION:
While functional balance metrics are increasingly being recognized as important objective indicators of disability associated with ASD, there is a need for a refinement of existing balance assessments to provide more clinically relevant information to better assist in the development of treatment strategies and in assessing treatment outcomes. The use of force plates and wearable sensors is growing among spine surgeons during patient assessments, so it is pertinent to refine test protocols that utilize this equipment rather than propose new methods with unproven or unfamiliar equipment. Standardization of a test protocol that utilizes existing technology to provide a more robust assessment of ASD patient balance performance will help spine surgeons better understand the characteristics of balance that are most affected by each patient's unique deformity and incorporate them into planning treatment strategies. Additionally, demonstration of the time requirements for this evaluation protocol is a critical step in establishing clinical relevance and efficacy for ASD patient care.

Data generated from this study will serve as important pilot data for additional studies focusing on the efficacy of the functional reach test to provide clinically relevant information on limits of functional balance among ASD patients. Information will provide guidance for both clinical decision-making and for objective techniques to assess postural balance of ASD patients.

The objectives of this research are as follows: 1) develop a clinically relevant protocol for assessing functional balance limits for ASD patients utilizing the functional reach test, 2) provide estimates of time requirements to conduct balance assessments in a spine clinic setting, and 3) provide preliminary data on postural balance limits of ASD patients and compare to them to matched asymptomatic controls.

ELIGIBILITY:
Adult Spinal Deformity Patient Inclusion Criteria:

* Adults over the age of 18
* Diagnosed with adult spinal deformity according to the SRS-Schwab Adult Spinal Deformity Classification System
* Indicated for deformity corrective surgery including multilevel spinal fusion of three or more levels
* Lowest instrumented level includes S1 or pelvic fixation
* Able to perform functional activities without the use of any assistance or support
* devices

Adult Spinal Deformity Patient Exclusion Criteria:

* Indicated for spinal fusion due to spinal tumor, trauma, or infection
* ASD patients who do not plan to be available for all follow-up evaluations at our institution
* Pregnancy during any time point within the participation duration

Asymptomatic Control Participant Inclusion Criteria:

* Adults over the age of 18
* No current or prior spine pathology or surgery
* Able to perform the functional activities without the use of any assistance or support devices

Asymptomatic Control Participant Exclusion Criteria:

* Any current or prior spine or lower extremity pathology or surgery that impacts the subject's ability to perform the functional activities
* Pregnancy at the time of the evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The adult spinal deformity (ASD) group will consist of adults with a diagnosis of scoliosis who are eligible for spinal deformity correcting surgery at the University of Kansas Medical Center.
  The asymptomatic control group will consist of adults who do not have any spinal diagnoses, have not have prior spinal fusions, and do not have any other conditions that affect their ability to perform the study activities.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Functional reach distance | Assessed preoperatively and at 3, 6, 12, and 24 month postoperative follow-ups
  The distance a participant can reach forward (in cm), to the side, and 45 degrees to the side with each arm
Center of pressure sway range | Assessed preoperatively and at 3, 6, 12, and 24 month postoperative follow-ups
  The range (in mm) that the participant's center of pressure moves in sagittal and coronal plane directions during the functional reach tests
Center of pressure velocity | Assessed preoperatively and at 3, 6, 12, and 24 month postoperative follow-ups
  The maximum and average velocity (in m/s) that the participant's center of pressure reaches during the functional reach tests
Center of pressure excursion | Assessed preoperatively and at 3, 6, 12, and 24 month postoperative follow-ups
  The summation of the distance (in mm) that the participant's center of pressure moves during the functional reach tests

SECONDARY OUTCOMES:
Patient reported pain level | Assessed preoperatively and at 3, 6, 12, and 24 month postoperative follow-ups
  Questionnaires assessing level of pain (0-10 on the numeric rating scale) for the mid-back, low-back, and both legs
Patient reported disability | Assessed preoperatively and at 3, 6, 12, and 24 month postoperative follow-ups
  A questionnaire called the Oswestry disability index (ODI) that assesses level of disability in performing activities of daily living
Timed up and go test | Assessed preoperatively and at 3, 6, 12, and 24 month postoperative follow-ups
  The time is takes to rise from a chair, walked forward 10 feet, turn around, and then sit back down

CONTACTS AND LOCATIONS:
Overall Officials: Damon Mar, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data from this study may be shared with other researchers in the future, but the type of data and the method of sharing has not been determined yet.